CLINICAL TRIAL: NCT07255976
Title: Comparison of Effectiveness of Gingival Displacement Using Retraction Cord and Aluminum Chloride Gel
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Armeen Fakhur, Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr Armeen Fakhur
Record Dates: First submitted 2025-11-19; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Gingival Bleeding; Prosthesis Failure, Dental; Tissue Injury
MeSH Terms: conditions — Gingival Hemorrhage; Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: In Group A, a knitted retraction cord (Ultra Pak, 0.00 mm) will be placed with a cord packer, and retraction gel applied using disposable syringe tips for 2 minutes. In Group B, gingival retraction gel with 25 % aluminum chloride (Ultradent) will be applied in the sulcus for 1-3 minutes, then rinsed with air-water spray. Impressions will be made by a one-step putty-light-body technique in metal trays, checked, disinfected, and poured with type II plaster. Casts will be coded separately. Time for placement of each system will be recorded with a stopwatch, haemorrhage control observed visually, and horizontal displacement measured by stereomicroscope and image analysis software at Dow Dental Lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retraction cord (Active Comparator): Conventionally used knitted cotton retraction cord
  Interventions: Device: knitted cotton retraction cord
- Aluminum chloride gel (Experimental): experimental 25% aluminum chloride gel retraction
  Interventions: Device: aluminum chloride gel

INTERVENTIONS:
Device: knitted cotton retraction cord — 00 size knitted cotton gingival displacement cord used as a control
  Other Names: conventional displacement cord
  Arms: Retraction cord
Device: aluminum chloride gel — 25% Aluminum chloride gel used as an experimental intervention
  Arms: Aluminum chloride gel

SUMMARY:
This study aims to compare the horizontal gingival displacement by using a retraction cord and aluminum chloride gel, and also to determine the time taken for placement and hemorrhage after the procedure by using a retraction cord and aluminum chloride gel. Patients of both genders, age ranges from 18 to 50 years, will be selecting requiring fixed prosthesis with of minimum two abutments. This study divided in two parallel groups of 33 patients in each group.

DETAILED DESCRIPTION:
To compare the effectiveness of a knitted retraction cord and 25% aluminum chloride-containing gel for horizontal gingival displacement, time taken for placement, patient discomfort and bleeding control after retraction cord removal and gel application with improved quality and better marginal fit of fixed prosthesis. This study include patients from range 18 to 50 years, Finishing line margins will be equigingival,Clinically and by radiographic analysis, healthy gingiva and periodontium around the abutments. Bleeding on probing index score-0 included,plaque index score(1-3) not included.

exclusion criteria is Sub-gingival or supra-gingival margins Patient having inappropriate root canal treated tooth. i.e Periapical pathosis over obturation, short root canal,Patient with probing depth 3mmm and above with uncontrolled bleeding. Patient with uncontrolled diabetes, hypertension or neurological disease.

SAMPLE TECHNIQUE: Non- probability consecutive sampling technique. Two groups will be formed among 66 patients with control group is retraction cord group and make two impressions after crown preparation with a finishing line Equiogingival margins will form than in group A in this study apply knitted retraction cord ultra Pak in thickness of .oo mm through retraction cord instrument by cord pecker retraction gel by company provided disposable tips with syringe into the circumferential area of sulcular preparation for 2 minutes and group B using gingival retraction gel containing 25% aluminum chloride viscous tat by ultra-dent after application of gingival retraction gel into sulcular area for 1-3minutes and wash with firm air water spray and will make impressions by one-step technique putty with the light body in metal stock trays then remove and check the impression for any inaccuracy then disinfect the impressions and pores with type 2 hard plaster and mention the code over cast that will not mix. The time required for placement of both gingival retraction systems will be recorded by using stopwatch in seconds and haemorrhage control will be checked by clinically observed with the naked eyes after air water spray up to 3 -5 seconds comparison of horizontal displacement on cast will be analyzed by stereomicroscope images using image analysis software at Dow dental lab.

ELIGIBILITY:
Inclusion Criteria:

1. age ranges from 18 to 50 years a fixed prosthesis with minimum of two abutments.
2. minimum of two abutments
3. Finishing line margins will be Equiogingival
4. Clinically healthy gingiva and periodontium.

Exclusion Criteria:

* 1. Sub-gingival or supra-gingival margins 2 Periapical pathosis 3. inadequate obturated root canals 4. bleeidng disorder 5.uncontrolled diabetes, 6.hypertension 7.neurological disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
horizontal gingival displacement | one time intervention , measure at baseline
  Horizontal displacement will be analyzed on casts using stereomicroscope imaging and image analysis software at Dow Dental Lab. and measurment in micron meter unit.

SECONDARY OUTCOMES:
placement time | one time intervention , measure at baseline
  time for placement will be recorded with a stopwatch.
bleeding control | one time intervention , measure at baseline
  bleeding control will be visual assist by after applying air-water spray.

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Fakhur, bds, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Armeen Fakhur, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No